CLINICAL TRIAL: NCT01633658
Title: The Variability of 25-hydroxyvitamin D Response From Crystalline 25-hydroxyvitamin D3 Compared to Native Vitamin D3: A Short Term Pharmacokinetic Study
Brief Title: The Variability of 25-hydroxyvitamin D Response From Crystalline 25-hydroxyvitamin D3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol has changed
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Creighton 13
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Cholecalciferol (Active Comparator): A single dose of 2500 micrograms cholecalciferol
  Interventions: Dietary Supplement: cholecalciferol
- 25(OH)D (Experimental): A single dose of 625 micrograms 25(OH)D
  Interventions: Dietary Supplement: 25(OH)D

INTERVENTIONS:
Dietary Supplement: cholecalciferol — a single dose of 2500 micrograms of cholecalciferol
  Arms: Vitamin D Cholecalciferol
Dietary Supplement: 25(OH)D — a single dose of 625 micrograms of 25(OH)D
  Arms: 25(OH)D

SUMMARY:
The investigators hypothesize that native vitamin D will have more variability in 25(OH)D dose response when compared to a given equipotent dose of 25-hydroxyvitamin D3. This will be a single blind, active control, pharmacokinetic study of 625 μg 25(OH)D given orally or 2500 μg native vitamin D given orally.

DETAILED DESCRIPTION:
Single blind, active control, pharmacokinetic study of 625 μg 25(OH)D given orally or 2500 μg native vitamin D given orally.

ELIGIBILITY:
Inclusion Criteria:

* Ten men and women in each group,
* aged 20-60.

Exclusion Criteria:

* History of hypercalcemia,
* vitamin D supplement use > 800 IU daily,
* BMI > 30,
* gastrointestinal malabsorption (from celiac sprue, colitis, surgery, etc.), kidney disease or liver disease,
* use of steroids in any form,
* anticonvulsants,
* antibiotics,
* acute illness, or
* vacation planned to "sunny climate"

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Serum 25(OH)D response | 28 days
  25(OH)D will be measured at frequent time intervals over 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armas, MD,MS, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States